CLINICAL TRIAL: NCT02621190
Title: Non-randomized Phase 2 Open-label Multicenter Study Determining the Response to Cabazitaxel in Metastatic Prostate Cancer (mCRPC) Patients With AR-V7 Positive Circulating Tumor Cells (CTCs): CARVE
Brief Title: Cabazitaxel in mCRPC Patients With AR-V7 Positive CTCs
Acronym: CARVE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no approval
Sponsor: Erasmus Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, M.P.J.K. Lolkema, oncologist, Erasmus Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL55865.078.15
Record Dates: First submitted 2015-11-24; First posted 2015-12-03 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Prostatic Neoplasms
Keywords: circulating tumor cells; predictive factor
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): patients without CTCs or AR-V7 negative CTCs are treated according to their physician's discretion
- B (Experimental): patients with AR-V7 positive CTCs are treated with cabazitaxel 25mg/m2 q3w
  Interventions: Drug: cabazitaxel

INTERVENTIONS:
Drug: cabazitaxel — 25mg/m2 q3w
  Other Names: Jevtana
  Arms: B

SUMMARY:
After failure on docetaxel, which has been the standard first line therapy for patients with metastatic castration-resistant prostate cancer (mCRPC), several treatment options are currently available. In retrospective studies, resistance has been described to two of the treatment options, enzalutamide and abiraterone, when a splice variant of the Androgen Receptor (AR-V7) is present on circulating tumor cells (CTCs). The investigators hypothesize that patients with AR-V7 positive CTCs do have a meaningful response to cabazitaxel.

DETAILED DESCRIPTION:
Rationale: After failure on docetaxel, which has been the standard first line therapy for patients with metastatic castration-resistant prostate cancer (mCRPC), several treatment options are currently available. Two of the treatment options are directed against the androgen receptor (AR), enzalutamide and abiraterone. A third option is cabazitaxel, a next generation taxane. No head-to-head comparisons have been done for these three therapies in second-line mCRPC and as of yet, the optimal choice is unknown. Resistance to the AR-targeted therapies is at least in part a consequence of signaling through constitutively active AR splice variants (AR-Vs).

Because AR splice variants only occur after conversion to a castration-resistant tumor, and can be acquired during systemic therapy for mCRPC, analysis of the castration-naïve primary tumor is not informative in the setting of second-line treatment of mCRPC. Circulating tumor cells (CTCs) can be analyzed repetitively and in real-time. Recently, AR-V7 mRNA expression in CTCs was shown to be associated with lack of response to AR-targeted therapy. AR-V7 mRNA expression does not seem to hinder response to cabazitaxel in the investigator's retrospective pilot study nor in a recently published small retrospective study.

Therefore the investigators hypothesize that the mRNA expression of AR-V7 in CTCs assessed before start of second-line treatment for mCRPC does not affect PSA response rate to cabazitaxel in patients who have progressed to docetaxel.

Objective: The primary objective of this study is to explore the PSA response rate to cabazitaxel in mCRPC patients who have progressed to docetaxel and have detectable AR-V7 expression in CTCs. Exploratory objectives include documenting the PSA response to cabazitaxel after enzalutamide or abiraterone treatment in initially AR-V7 negative patients, describing the toxicity of cabazitaxel in second and third-line treatment as well as exploring if response measured by CTC counts and PSA is related to systemic cabazitaxel exposure.

Study design: This is a multicenter, non-randomized phase 2 study. Patients will be allocated to one of the following treatment groups according to the results of CTC enumeration and characterization in the screening phase:

Group A: Patients with <3 CTCs and patients with ≥3 CTCs without AR-V7 expression will receive physician's choice of treatment Group B: Patients with ≥3 CTCs with AR-V7 expression will receive Cabazitaxel 25 mg/m² every 3 weeks plus prednisone 10 mg daily.

Patients in group A who are treated with enzalutamide or abiraterone and experience disease progression, can then again enter the screening phase and, after additional eligibility check, subsequently be treated with cabazitaxel in group B if ≥3 CTCs are present and AR-V7 mRNA expression is now detected. These patients will not be re-included in the study.

Study population: Adult mCRPC patients, age≥18 years, who progressed during docetaxel treatment. Prior enzalutamide or abiraterone treatment is permitted.

Intervention: In all patients, 2 x 10 mL blood will be drawn for enumeration and isolation of CTCs at baseline. In group B, cabazitaxel will be administrated intravenously at a dose of 25 mg/m², during a one-hour infusion every 3 weeks, as well as continuous treatment with prednisone 5 mg orally twice daily, or 10 mg once daily, according to standard care. In these patients, an additional 2 x 10 mL blood will be drawn after the second cycle of treatment for CTC enumeration and isolation. In group B, an additional 10 mL blood will be drawn for storage of plasma at baseline and before start of every every cycle (i.e., every 3 weeks) for analysis of cell-free DNA (cfDNA) as part of a side-study. In group B, also 4 x 5 mL blood (baseline; end of infusion, 2 and 6 hours after end of the first cabazitaxel infusion) will be drawn for a pharmacokinetic side-study, to explore a cabazitaxel exposure effect relation. Patients in group A will be treated according to their physician's choice. In group A, an additional 10 mL blood will be drawn for storage of plasma at baseline, at 12 weeks after start of treatment and upon progression to enzalutamide or abiraterone for analyses of cell-free DNA (cfDNA) as part of a side-study. Patients in group A who receive abiraterone or enzalutamide and subsequently experience disease progression can again enter the screening phase of the study, and if eligible, be included in group B.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

For the CTC enumeration and isolation, a total of 40 mL additional blood will be drawn at the time of regular blood draws (treatment group A: 1 x 20 mL at baseline and 1 x 20 mL upon progression to enzalutamide or abiraterone; treatment group B: 1 x 20 mL at baseline and 1 x 20 mL after the second cycle of cabazitaxel).

For storage of plasma for cfDNA analysis, a total of 100 mL additional blood will be drawn at the time of regular blood draws (at baseline and before each treatment cycle) from patients in group B. In group A, for storage of plasma for cfDNA analysis, a total of 30 mL additional blood will be drawn at the time of regular blood draws (at baseline, at 12 weeks after start of treatment and upon disease progression).

For pharmacokinetic analysis, in patients in group B, a total of 20 mL (4 x 5 mL) additional blood will be drawn at baseline, end of infusion, 2 and 6 hours after the first cabazitaxel infusion.

Cabazitaxel is standard second-line chemotherapy for mCRPC patients. In the TROPIC trial, the most common observed grade 3-4 toxicity was neutropenia (82%). Despite the high incidence of neutropenia, febrile neutropenia was rare (8%). The most frequent non-hematologic adverse event (AE) was diarrhea, occurring in 47% (grade ≥3 6%) of patients treated with cabazitaxel, compared to 11% (grade ≥3 <1%) of patients treated with mitoxantrone. In the TROPIC trial, a total of 18 (5%) patients treated with cabazitaxel died within 1 month of the last drug infusion due to adverse effects. This compares to 3 drug-related deaths (2%) in the mitoxantrone group. The most common cause of death in patients treated with cabazitaxel was neutropenia and its clinical consequences. The frequency of hematological adverse events and related deaths demonstrates that cabazitaxel treatment requires careful monitoring and management of emerging symptoms. Dose reductions as well as supportive treatment (i.e. the administration of granulocyte colony-stimulating factor [G-CSF]) will be considered to manage the toxic effects of treatment.

Patients in group B will have scheduled study visits frequently, in accordance with standard-of-care cabazitaxel treatment. Patients will return for regularly scheduled study visits for as long as they continue study treatment, or discontinued study treatment but have not yet experienced disease progression. All patients will be followed for survival after discontinuing treatment. For the primary endpoint, serial blood samples will be collected every three weeks to quantify PSA. Radiographic evaluations (bone scans and CT/MRI-scans of the abdomen and pelvis) will be employed after four and eight cycles of cabazitaxel to assess the status of the disease according to modified RECIST 1.1 criteria.

The safety of cabazitaxel in second and third-line treatment will be assessed by monitoring the frequency of treatment related (serious) adverse events, which will be recorded according to the Common Terminology Criteria (CTCAE) scale version 4.03.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features.

  * Continued androgen deprivation therapy either by LHRH agonists/antagonists or orchiectomy.
  * Serum testosterone <50 ng/mL (1.7 nmol/L) within 21 days before treatment group allocation.
  * Age ≥18 years
  * Disease progression during or after treatment with docetaxel. Disease progression for study entry is defined as one or more of the following criteria:

    * PSA progression defined by at least 2 consecutive PSA rises over a reference value, with an interval of ≥ 1 week between each determination. PSA at screening visit should be ≥ 2.0 μg/l.
    * Bone disease progression defined by the appearance of new lesions on a bone scan, confirmed on a second bone scan ≥ 6 weeks later.
    * Soft tissue disease progression defined by modified RECIST criteria 1.1 (baseline LN size must be ≥ 2.0 cm to be considered target or evaluable lesion) (15)
  * ECOG performance status 0-2 (appendix A)
  * Written informed consent according to ICH-GCP before study treatment and any study specific procedures

Exclusion Criteria:

* Impossibility or unwillingness to take oral drugs

  * Geographical, psychological or other non-medical conditions interfering with follow-up
  * Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus or active systemic or local bacterial, viral, fungal - or yeast infection)
  * Symptomatic CNS metastases or history of psychiatric disorder that would prohibit the understanding and giving of informed consent.
  * Chemotherapy or immunotherapy (other than LHRH analogues) within the last 4 weeks before study inclusion.
  * Prior treatment with cabazitaxel
  * Successive treatment with both abiraterone and enzalutamide in the post-docetaxel setting
  * Radiotherapy to 40% or more of the bone marrow
  * Known hypersensitivity to corticosteroids
  * History of severe hypersensitivity reaction (≥grade 3) to docetaxel
  * History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs
  * Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments) (see Appendix C)
  * Concomitant vaccination with yellow fever vaccine
  * Abnormal liver functions consisting of any of the following (within 21 days before treatment group allocation):
  * Total bilirubin > 1.5 x ULN (except for patients with documented Gilbert's disease)
  * If total bilirubin > 1 x ULN or AST > 1.5 x ULN inclusion is permitted but cabazitaxel dose should be reduced 20mg/m2
  * Abnormal hematological blood counts consisting of any of the following (within 21 days before treatment group allocation):
  * Absolute neutrophil count < 1.5 x 109/L
  * Platelets < 100 x 109/L
  * Hemoglobin < 6.2 mmol/L

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Prostate specific antigen (PSA) response rate | 12 weeks after start of treatment
  PSA response rate is defined as a reduction of at least 50% from baseline during therapy, confirmed after ≥4 weeks by an additional PSA evaluation.

SECONDARY OUTCOMES:
Circulating tumor cell (CTC) response rate | 9 weeks after start of treatment
  CTC Response rate is defined as a decrease from ≥5 CTCs per 7.5 mL blood at baseline to <5 CTCs per 7.5 mL blood, as measured by the CellSearch system
Prostate specific antigen (PSA) change from baseline | 12 weeks after start of treatment
  • PSA change from baseline at 12 weeks defined as the percent change in PSA from baseline (rise or fall) at 12 weeks, according to PCWG2 criteria.
Maximum Prostate specific antigen (PSA) decrease | through study completion, an average of two years
  Maximum PSA decrease is defined according to PCWG2 criteria (30), i.e., the maximal change (rise or fall) at any time through study completion, illustrated by a waterfall plot
Progression-free survival | from date of treatment allocation until the date of first documented progression (see description) or date of death from any cause, whichever came first, assessed through study completion, up to 100 months
  Progression defined as:
  * At least 2 consecutive PSA rises over a reference value, with an interval of ≥ 1 week between each determination. PSA at screening visit should be ≥ 2.0 μg/l; the date of progression will be the first of the 2 consecutive dates.
  * Soft tissue disease progression defined by modified RECIST criteria (1.1) (baseline LN size must be ≥ 2.0 cm to be considered target or evaluable lesion).
  * Bone disease progression defined by the appearance of new lesions on a bone scan, confirmed on a second bone scan ≥ 6 weeks later. Ambiguous results should be confirmed by other imaging modalities (e.g., CT or MRI). The date of progression will be the first of the 2 consecutive dates.
Overall survival | time from treatment group allocation to death due to any cause, assessed through study completion, up to 100 months
grade 3-4 adverse events and serious adverse events (SAEs) | through study treatment until 30 days after end of treatment
Cabazitaxel concentration in the blood (measured in ng/mL) | during the first cycle of cabazitaxel, until 6 hours after end of cabazitaxel infusion
Total systemic exposure to cabazitaxel (measured in mg/m2) | through study treatment, an average of 10 cycles, i.e., 30 weeks of treatment
AR-V7 mRNA expression as well as mRNA expression of other splice variants in CTCs indicated as absent (-) or present (+) on a per-patient basis | at screening visit

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC Cancer Institute, Rotterdam, Netherlands